CLINICAL TRIAL: NCT03448575
Title: A Targeted Approach To A Safer Use of Antipsychotics In Youth
Brief Title: Safer Use of Antipsychotics in Youth
Acronym: SUAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Nationwide Children's Hospital (Other); Seattle Children's Hospital (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HHSN271201600002C
Record Dates: First submitted 2018-02-21; First posted 2018-02-28 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Child Behavior Disorders
Keywords: Youth; Mental Health; Psychotropic; Medication Safety; Quality Improvement
MeSH Terms: conditions — Child Behavior Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Providers are preassigned to one of two study arms: usual care control or intervention arm. Patients are assigned to the same arm as the provider triggering the best practice alert and study algorithm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Waivers of consent have been obtained for providers and for patients/parents/guardians. None are informed of the study design or study activities by arm. The investigator is blind to study arm assignment of providers and patients. Only automated data collection is utilized for this practical trial. Study arm is masked for the programmer/analyst pulling outcomes data from health system records. Study arm will also be masked for study staff verifying study eligibility prior to the official study enrollment. Arm is not masked for study intervention staff (consulting psychiatrists, behavioral health navigators, bridging therapists) since these staff only interact with intervention arm subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Medication Alert Only (Sham Comparator): The control arm medication alert is a simple text pop-up in the EMR that will inform the prescriber of Choosing Wisely® recommendations developed the American Psychiatric Association regarding antipsychotic medication use in children and adolescents.
  Interventions: Other: Control - Provider Medication Alert Only
- Intervention - Alert + CAP Review AND Enhanced BH Access (Experimental): The intervention alert prompts the prescriber to keep/remove the antipsychotic order, and/or order any study services: behavioral health navigation, expedited psychotherapy access, virtual consult with a child and adolescent psychiatrist (CAP). Passive case review by the study CAP will occur for all intervention arm cases. A virtual consult will be scheduled if the prescriber ordered it or the CAP needs to discuss the case. The CAP will provide the prescriber with a written summary of his/her review.
  Following review by the CAP, a navigator reaches out to the eligible intervention arm patient/family to offer extra support. The navigator's role is to (a) provide extra support to facilitate access and engagement in appropriate psychosocial therapies; (b) coordinate short-duration bridging therapy sessions for teens/families not engaged in psychotherapy, when appropriate; and (c) keep the prescriber informed of any clinically relevant updates.
  Interventions: Other: Intervention - Alert + CAP Review AND Enhanced BH Access

INTERVENTIONS:
Other: Control - Provider Medication Alert Only — Simple text medication alert referencing Choosing Wisely guidelines.
  Arms: Control - Medication Alert Only
Other: Intervention - Alert + CAP Review AND Enhanced BH Access — Interactive medication alert referencing SUAY Clinical Guidelines and offering options to keep/remove orders for the antipsychotic, virtual CAP consult, BH navigation for the patient, and access to bridging therapy for the patient.
  Arms: Intervention - Alert + CAP Review AND Enhanced BH Access

SUMMARY:
This study tests the effectiveness of an intervention treatment algorithm vs. usual care control in a practical clinical trial. Control arm providers will receive a standard medication alert in the electronic medical record (EMR) when initiating an antipsychotic prescription for an eligible patient. Intervention arm prescribers will receive an interactive medication alert in the EMR when prescribing for eligible patients and the patient and provider will enter the treatment algorithm (provider - medication alert plus clinical review by a child psychiatrist; patient - offer of personalized behavioral health navigation plus bridging therapy when appropriate). The study aims to recruit 800 eligible patients in 4 health systems.

DETAILED DESCRIPTION:
SUAY is a practical clinical trial designed to test the effectiveness of an intervention aiming to improve the targeted and safer use of antipsychotic medications by guiding clinician-prescribing behavior of antipsychotics for children aged ≥ 3 and < 18 years and encouraging psychosocial therapy for eligible youth. The intervention includes a medication best practice alert in Epic, consultation with a child and adolescent psychiatrist, and extra support for patients and families to improve behavioral health service access. The trial will be conducted in 4 non-academic health systems. Each health system will randomize prescribers to one of two study arms, intervention and control. During patient encounters, entering an antipsychotic for a potentially eligible patient will cause either the control or intervention medication alert to fire in the electronic medical record. The control arm medication alert will point prescribing clinicians to relevant Choosing Wisely® recommendations. The intervention arm medication alert will inform prescribers that:

1. Antipsychotics are not recommended 1st line treatment for non-psychotic disorders;
2. A child and adolescent psychiatrist (CAP) will review antipsychotic usage by youth;
3. Expedited access to bridging therapy, behavior health navigation, and/or a proactive consultation with a CAP may be ordered.

The intervention medication alert will point prescribing clinicians to both Choosing Wisely® recommendations and to SUAY clinical prescribing guidelines. SUAY guidelines were developed by a national expert consensus panel in a prior phase of the study.

Analytic data will be collected from automated data sources at the health systems. The primary outcomes are percent of children ordered an antipsychotic medication at 6 months of follow up, and total person-months of antipsychotic orders placed for participants during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 3 and < 18 years of age at the time of the encounter at which the study alert fired (index date);
* Patient is initiating a new episode of outpatient treatment with an antipsychotic medication. (New episodes are defined by no record of an antipsychotic medication being ordered within the health system as part of an outpatient care plan in the prior 180 days);
* Study service (BH navigation, bridging therapy, CAP consult) ordered in Epic for the patient; (e.g., provider removed antipsychotic order and still ordered study services);

Exclusion Criteria:

* Patient has a diagnosed psychotic disorder, mania, autism spectrum disorder, or intellectual disability;
* Patient was enrolled in the SUAY pilot study;
* The antipsychotic entered is prochlorperazine (Comazol®);
* An outpatient antipsychotic order is entered by a temporary provider in the health system (e.g., "doc of the day"). Orders placed by temporary providers do not count towards the 180 day medication free period for defining a new episode of care.
* The antipsychotic order was placed within an urgent care, emergency department, or inpatient setting (to avoid intervening during a crisis). Orders placed in these settings do not count towards the 180 day medication free period for defining a new episode of care.
* Primary language is not English

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 733 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Penfold, PhD, Principal Investigator — Kaiser Permanente
Locations (4):
- United States (4):
  - Kaiser Permanente Colorado Institute for Health Research, Aurora, Colorado
  - Nationwide Children's Hospital / Partners for Kids, Columbus, Ohio
  - Kaiser Permanente Center for Health Research - Northwest, Portland, Oregon
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The data sharing plan is incorporated by reference into the contract governing the project. Any changes to the plan must be pre-approved by the NIH Contracting Officer. A de-identified database will be delivered to the NIH, along with a statistical report. Any datasets for public distribution (including to the National Database for Clinical Trials Related to Mental Illness) will be de-identified in compliance with HIPAA standard for de-identification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: A de-identified database will be delivered to the NIH on or before 12/24/2021, along with data dictionary and a study report.
Access Criteria: Access to contact deliverables will be determined by NIH.

REFERENCES:
- [Derived] Chavez LJ, Richards JE, Fishman P, Yeung K, Renz A, Quintana LM, Massimino S, Penfold RB. Cost of Implementing an Evidence-Based Intervention to Support Safer Use of Antipsychotics in Youth. Adm Policy Ment Health. 2023 Sep;50(5):725-733. doi: 10.1007/s10488-023-01273-y. Epub 2023 Jun 1. PMID 37261566
- [Derived] Penfold RB, Thompson EE, Hilt RJ, Schwartz N, Robb AS, Correll CU, Newton D, Rogalski K, Earls MF, Kowatch RA, Beck A, Yarborough BJH, Crystal S, Vitiello B, Kelleher KJ, Simon GE. Development of a Symptom-Focused Model to Guide the Prescribing of Antipsychotics in Children and Adolescents: Results of the First Phase of the Safer Use of Antipsychotics in Youth (SUAY) Clinical Trial. J Am Acad Child Adolesc Psychiatry. 2022 Jan;61(1):93-102. doi: 10.1016/j.jaac.2021.04.010. Epub 2021 May 4. PMID 34256967
- [Derived] Chavez LJ, Kelleher KJ, Beck A, Clarke GN, Penfold RB. Trends Over Time in Antipsychotic Initiation at a Large Children's Health Care System. J Child Adolesc Psychopharmacol. 2021 Jun;31(5):381-386. doi: 10.1089/cap.2020.0190. PMID 34143677
- [Derived] Penfold RB, Thompson EE, Hilt RJ, Kelleher KJ, Schwartz N, Beck A, Clarke GN, Ralston JD, Hartzler AL, Coley RY, Akosile M, Vitiello B, Simon GE. Safer use of antipsychotics in youth (SUAY) pragmatic trial protocol. Contemp Clin Trials. 2020 Dec;99:106184. doi: 10.1016/j.cct.2020.106184. Epub 2020 Oct 20. PMID 33091587
- [Derived] Schoenfelder Gonzalez E, Myers K, Thompson EE, King DA, Glass AM, Penfold RB. Developing home-based telemental health services for youth: Practices from the SUAY Study. J Telemed Telecare. 2021 Feb;27(2):110-115. doi: 10.1177/1357633X19863208. Epub 2019 Jul 25. PMID 31342851

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We define "started" as the number of eligible participants for whom a study medication alert fired in Epic when the provider ordered an antipsychotic. A blinded study team member assessed for eligibility according to study criteria and marked as eligible or ineligible.
Groups:
- Intervention - Alert + CAP Review AND Enhanced BH Access: The intervention alert prompts the prescriber to keep/remove the antipsychotic order, and/or order any study services: behavioral health navigation, expedited psychotherapy access, virtual consult with a child and adolescent psychiatrist (CAP). Passive case review by the study CAP will occur for all intervention arm cases. A virtual consult will be scheduled if the prescriber ordered it or the CAP needs to discuss the case. The CAP will provide the prescriber with a written summary of his/her review.
  Following review by the CAP, a navigator reaches out to the eligible intervention arm patient/family to offer extra support. The navigator's role is to (a) provide extra support to facilitate access and engagement in appropriate psychosocial therapies; (b) coordinate short-duration bridging therapy sessions for teens/families not engaged in psychotherapy, when appropriate; and (c) keep the prescriber informed of any clinically relevant updates.
  Intervention - Alert + CAP Review AND Enhanced BH Access: Interactive medication alert referencing SUAY Clinical Guidelines and offering options to keep/remove orders for the antipsychotic, virtual CAP consult, BH navigation for the patient, and access to bridging therapy for the patient.
Period: Overall Study
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access
Started | 385 | 348
Completed | 385 | 348
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access | Total
Number analyzed (Participants) | 385 | 348 | 733
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 385 | 348 | 733
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 183 | 366
  Male | 202 | 165 | 367
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 22 | 40
  Not Hispanic or Latino | 324 | 283 | 607
  Unknown or Not Reported | 43 | 43 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 35 | 29 | 64
  White | 282 | 265 | 547
  More than one race | 33 | 23 | 56
  Unknown or Not Reported | 30 | 25 | 55
Region of Enrollment [Number; unit: participants]
  United States | 385 | 348 | 733

OUTCOME MEASURES:

1. Primary Outcome: Percent of Youths With Antipsychotic Orders at 6 Months
Description: Measured by medication orders placed within the health system
Time Frame: 180 day period following index date
Measure: Number; unit: percentage of youths
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access
Number analyzed (Participants) | 385 | 348
percentage of youths | 54.6 | 47.6

2. Primary Outcome: Days' Supply of Antipsychotics Ordered for Youth
Description: Average days' supply of antipsychotic medication (values fell between 1 and 180 days), as measured by the intended days' supply on the medication orders for each participant. Only orders placed within the health system were accounted for.
Time Frame: 180 day period following index date
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access
Number analyzed (Participants) | 385 | 348
days | 128.2 (57.9) | 118.5 (61.6)

3. Secondary Outcome: Percent of Youths Using Antipsychotics at 6 Months
Description: Measured by medication fill data available to the health system
Time Frame: 180 day period following index date
Measure: Number; unit: percent of youths
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access
Number analyzed (Participants) | 385 | 348
percent of youths | 39.1 | 35.5

4. Secondary Outcome: Days' Supply of Antipsychotic Use by Youth
Description: Average days' supply of antipsychotic medication (values fell between 1 and 180 days), as measured by medication fill data available to the health system for each participant. Only pharmacy claims captured by the health system were accounted for.
Time Frame: 180 day period following index date
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access
Number analyzed (Participants) | 385 | 348
days | 95.2 (62.0) | 87.7 (60.5)

5. Secondary Outcome: Emergency Department/Urgent Care Visit Frequency
Description: Measured by utilization data; both for psychiatric crises and for all other reasons
Time Frame: 180 day period following index date
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access
Number analyzed (Participants) | 385 | 348
number of visits | 0.43 (0.98) | 0.36 (0.99)

6. Secondary Outcome: Baseline and Follow-up Safety Assessments - BMI
Description: Percentage of patients with BMI measurements completed at baseline and 3 months
Time Frame: index date to 180 days post-index date
Measure: Number; unit: percent of patients
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access
Number analyzed (Participants) | 385 | 348
percent of patients | 65.5 | 54.9

7. Secondary Outcome: Change to Psychotropic Medication Treatment Plan
Description: Percentage of patients with change to psychotropic medication treatment plan following exposure to study algorithm
Time Frame: 180 day period following index date
Measure: Number; unit: percent of patients
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access
Number analyzed (Participants) | 385 | 348
percent of patients | 42.3 | 40.8

8. Secondary Outcome: Behavioral Health (BH) Navigation Acceptance
Description: Percent of intervention arm patients that agree to BH navigation
Time Frame: 180 day period following index date
Population: Control arm patients were not offered behavioral health navigation.
Measure: Number; unit: percent of patients
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access
Number analyzed (Participants) | 0 | 348
percent of patients |  | 55.5

9. Secondary Outcome: Use of Usual Care Therapy
Description: Percentage of patients attending two or more system-provided therapy sessions
Time Frame: 180 day period following index date
Measure: Number; unit: percentage of patients
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access
Number analyzed (Participants) | 385 | 348
percentage of patients | 47.3 | 53.5

10. Secondary Outcome: Use of Bridging Therapy
Description: Percentage of patients attending two or more study-provided bridging therapy sessions
Time Frame: 180 day period following index date
Population: Control arm patients were not offered bridging therapy.
Measure: Number; unit: percent of patients
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access
Number analyzed (Participants) | 0 | 348
percent of patients |  | 1.4

11. Secondary Outcome: Use of Usual Care Therapy Following Bridging Therapy
Description: Of patients in study therapy, percentage who subsequently attend two or more system-provided therapy sessions
Time Frame: 180 day period following index date
Population: Formal statistical analyses were not conducted because only 5 intervention participants elected to participate in bridging therapy, which is too few participants to measure differences in subsequent use of usual care. Bridging therapy was not offered to control participants.
Measure: Number; unit: percent of patients
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access
Number analyzed (Participants) | 0 | 348
percent of patients |  | 1.437

12. Secondary Outcome: Baseline and Follow-up Safety Assessments - Safety Lab Tests
Description: Percentage of patients with safety lab tests ordered and completed at baseline and 3 months
Time Frame: index date to 180 days post-index date
Measure: Number; unit: percent
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access
Number analyzed (Participants) | 385 | 348
percent | 32.5 | 28.2

ADVERSE EVENTS:
Time Frame: 6 months per individual over a 2.5 year study period
Description: No difference
Arm/Group | Control - Medication Alert Only | Intervention - Alert + CAP Review AND Enhanced BH Access
All-Cause Mortality (participants affected / at risk) | 0/385 | 0/348
Serious Adverse Events (participants affected / at risk) | 0/385 | 0/348
Other Adverse Events (participants affected / at risk) | 0/385 | 0/348

LIMITATIONS AND CAVEATS:
While inclusion/exclusion criteria were manually confirmed by chart review, ~7% of patients enrolled with an exclusion diagnosis. We obtained this information via administrative claims data at study end. External claims data were unavailable in real time when the BPA fired.

EHR functionality cannot differentiate a de novo prescription order from a "historical medication". Some new patients had initial prescriptions written elsewhere; the BPA fired when study clinicians continued treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT03448575/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT03448575/SAP_001.pdf